CLINICAL TRIAL: NCT03306550
Title: Research on Mechanism of Drug-drug Interaction Between Salvianolate Injection and Aspirin Based on the Metabolic Enzyme and PK-PD Model
Brief Title: Mechanism of Drug-drug Interaction Between Salvianolate Injection and Aspirin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zz0908022
Record Dates: First submitted 2017-09-04; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-08

CONDITIONS: Angina, Stable
Keywords: drug-drug interaction; Asprin; salvianolate injection; PK-PD model; metabolic enzymes
MeSH Terms: conditions — Angina, Stable | interventions — salvianolate; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aspirin arm (Active Comparator): only take aspirin (100mg,qd) orally for 10 days treatment course
  Interventions: Drug: Aspirin Tablet
- salvianolate injection arm (Active Comparator): only inject salvianolate(200mg+5%Glucose Injection 250ml，iv) for 10 days treatment course
  Interventions: Drug: salvianolate injection
- aspirin and salvianolate injection arm (Experimental): take aspirin (100mg,qd) orally and inject salvianolate(200mg+5%Glucose Injection 250ml，iv) for 10 days treatment course
  Interventions: Drug: salvianolate injection; Drug: Aspirin Tablet

INTERVENTIONS:
Drug: salvianolate injection — The main ingredient of salvianolate injection is salvianolic acid B(SAB) which is extracted from the root of red salvia. Red salvia is used in traditional Chinese Medicine. It could promote blood circulation to removing blood stasis,which is clinically effective in treatment for cardiovascular disease.
  Arms: aspirin and salvianolate injection arm; salvianolate injection arm
Drug: Aspirin Tablet — Anti-platelet medicine treatment and Chinese traditional medicine (TCM) promoting blood circulation to removing blood stasis is widely used in treatment for cardiovascular disease.
  Arms: aspirin and salvianolate injection arm; aspirin arm

SUMMARY:
The combination of anti-platelet medicine treatment and Chinese traditional medicine (TCM) promoting blood circulation to removing blood stasis is widely used in treatment for cardiovascular disease. However, the material foundation, effective mechanism and drug-drug interaction is still not clear. In order to solve the puzzle of rational use of Joint application by TCM and Western Medicine(WM),investigators conduct a research on mechanism of drug-drug interaction between salvianolate injection and aspirin based on metabolic enzyme and PK-PD model. This clinical trial contain three groups, aspirin group, salvianolate injection group and combination (salvianolate injection+aspirin) group. Investigators collect blood samples at special time points during post-administration.Investigators have already find out the Salvianolate's pharmacokinetic characteristics in vivo and establish the biological sample-testing analysis method in previous research. Depending on these results, this clinical trial aim to explore the pharmacodynamics-pharmacokinetics(PK-PD) characteristics of combination with Salvianolate and aspirin through biomarkers, blood concentration. Finally clarify the TCM and WM material basis and mutual mechanism of drug interaction and guide reasonable clinical prescription.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of coronary heart disease.
2. Meet the diagnostic criteria of stable angina pectoris.
3. Meet the diagnostic criteria of syndrome of blood stasis.
4. Angina in grade I-II according to Canadian cardiovascular society (CCS).
5. It could be enrolled if the subject taking aspirin or salvianolate injection with one month regularly。
6. The subjects were informed and voluntarily signed informed consent.

Exclusion Criteria:

1. Severe heart disease (acute myocardial infarction of acute myocardial infarction in 6 months), severe cardiopulmonary dysfunction (eg: cardiac function II)
2. Poorly controlled hypertension(systolic pressure >160mmHg or diastolic pressure >100mmHg).
3. Diabetics.
4. Severe primary diseases such as liver and renal hematopoietic system damage. Such as:liver function（ALT≥2×ULN、AST≥2×ULN）,kidney function（Cr>1.0×ULN) or nervous and mental disorder.
5. Pregnant, breast-feeding and menstrual women, or women planning pregnancy within 3 months.
6. Subjects who participated in clinical trials in recent 3 months.
7. Subjects who took surgery treatment or had hemorrhagic tendency in recent 4 weeks.
8. Subjects who had drug allergy history or with allergic constitution.
9. Subjects who has mental or physical disorders.
10. Subjects who had bad compliance or is not suitable for this clinical trial by investigator's judgement

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-10-10 (Estimated); Primary Completion 2018-04-10 (Estimated); Study Completion 2018-10-10 (Estimated)

PRIMARY OUTCOMES:
Change of P-selection expression(platelet activation-dependent granule membrane) at different time points. | Getting blood sample before taking medicine in the day 10 and after it in 15min、1h、2h、8h、24h
  Use flow cytometric method to detect the P-selection expression on platelet at different time points. Analyse the influence of Asprin/Salvianolate on platelet interaction adhesion during drug concentration-time curves.
Change of PAC-1 expression (platelet-associated complement) on the activated platelets at different time points. | Getting blood sample before taking medicine in the day 10 and after it in 15min、1h、2h、8h、24h
  Use flow cytometric method to detect the PAC-1 expression on platelet at different time points. Analyse the influence of Asprin/Salvianolate on platelet aggregation during drug concentration-time curves.
Change of P2Y12 acceptor expression on platelets at different time points. (P2Y12 acceptor is a receptor for ADP(adenosine diphosphate) and ATP (adenosine triphosphate )coupled to G-proteins that inhibit the adenylyl cyclase second messenger system) | Getting blood sample before taking medicine in the day 10 and after it in 15min、1h、2h、8h、24h
  Use flow cytometric method to detect the P2Y12 acceptor expression on platelet at different time points. Analyse the influence of Asprin/Salvianolate on platelets aggregation activated by ADP or ATP during drug concentration-time curves.
Change of PDE enzymes（phosphodiesterase）expression on platelet at different time points. | Getting blood sample before taking medicine in the day 10 and after it in 15min、1h、2h、8h、24h
  Use ELISA method to detect the PDE enzymes expression at different time points. Analyse the influence of Asprin/Salvianolate on platelets activated by PDE enzymes during drug concentration-time curves.

SECONDARY OUTCOMES:
Change of Aspirin esterase activity at different blood concentration of Asprin/Salvianolate | Getting blood sample before taking aspirin in day 8 and day 9.In the day 10, getting blood sample before taking aspirin and after taking aspirin in 5min、15min、30min、45min、1h、2h、4h、8h、12h、24h
  Conduct biological analysis by LC-MS/MS(liquid chromatography tandem mass spectrometry) to detect Aspirin and salicylic aspirin and salicylic acid:CSA/C(ASA+SA).The activity of combination arm and of the asprin arm is compared by t test.
Change of Catechol-o-methyltransferase (COMT) activity at different blood concentration of Asprin/Salvianolate | Getting blood sample before injection in day 8 and day 9.In the day 10, getting blood sample before injection and after injection in 5min、15min、30min、45min、1h、2h、4h、8h、12h、24h
  COMT activity is the main metabolic enzymes of SAB.Use kit to detect COMT activity .

REFERENCES:
- [Derived] Cao W, Yang Q, Zhang W, Xu Y, Wang S, Wu Y, Zhao Y, Guo Z, Li R, Gao R. Drug-drug interactions between salvianolate injection and aspirin based on their metabolic enzymes. Biomed Pharmacother. 2021 Mar;135:111203. doi: 10.1016/j.biopha.2020.111203. Epub 2021 Jan 3. PMID 33401223
- [Derived] Zhang W, Zhu B, Cao W, Li R, Wang S, Gao R. Research on the mechanism of drug-drug interaction between salvianolate injection and aspirin based on the metabolic enzyme and PK-PD model: study protocol for a PK-PD trial. Trials. 2018 Sep 14;19(1):491. doi: 10.1186/s13063-018-2861-7. PMID 30217228